CLINICAL TRIAL: NCT03075254
Title: Central Mechanisms of Chronic Pain and Fatigue Subtitle: Functional Imaging of Brain and Spinal Cord
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201602417 -N-A
Record Dates: First submitted 2017-02-23; First posted 2017-03-09 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Chronic Fatigue Syndrome; Fibromyalgia
Keywords: Pain; Fatigue
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Fibromyalgia; Pain; Fatigue | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Healthy Control: normal volunteers (HC) Undergoing sensory testing, brain and spinal cord neuroimaging and Inventory assessments.
  Interventions: Device: A Peltier for Sensory testing; Device: functional magnetic resonance imaging for Brain Neuroimaging; Device: fMRI for Spinal Cord Neuroimaging
- Fibromyalgia Only: The diagnosis of FM will require a history of chronic widespread pain as well as the presence of at least eleven out of eighteen paired tender points. Undergoing sensory testing, brain and spinal cord neuroimaging and Inventory assessments.
  Interventions: Device: A Peltier for Sensory testing; Device: functional magnetic resonance imaging for Brain Neuroimaging; Device: fMRI for Spinal Cord Neuroimaging
- Chronic fatigue and Fibromyalgia Syndrome: Diagnosis of ME/CFS will require a history of chronic fatigue persisting or relapsing for more than 6 months as well as the presence of at least four out of eight designated symptoms. Undergoing sensory testing, brain and spinal cord neuroimaging and Inventory assessments.
  Interventions: Device: A Peltier for Sensory testing; Device: functional magnetic resonance imaging for Brain Neuroimaging; Device: fMRI for Spinal Cord Neuroimaging

INTERVENTIONS:
Device: A Peltier for Sensory testing — Subjects will be trained to rate the magnitude of late sensations elicited following brief (700 msec) contact of a preheated thermode with the glabrous (palmar) skin of either hand/foot either numerically or using a visual analogue scale.
  Other Names: Heat Foil device
Device: functional magnetic resonance imaging for Brain Neuroimaging — to evaluate baseline changes in regional cerebral blood flow to nociceptive thermal stimuli applied to the extremities of FM patients and healthy volunteers.
  Other Names: fMRI
Device: fMRI for Spinal Cord Neuroimaging — The subjects will be positioned supine and immobilized by means of a padded head support. The spinous process of the first thoracic vertebra (T1) will be aligned with the center of surface Neuro - coil. This coil will be employed for both transmission of radio-frequency (RF) pulses and detection of the magnetic resonance (MR) signal. A modified FLASH sequence will be employed to obtain Blood Oxygen Level Dependent (BOLD)-sensitive images of the spinal cord.
  Other Names: functional magnetic resonance imaging

SUMMARY:
Chronic pain and fatigue are characterized by peripheral and central mechanisms including low pain thresholds, temporal summation, peripheral and central sensitization. This application will focus on central factors of chronic pain and fatigue. Functional brain imaging will be used to characterized brain and spinal cord abnormalities that contribute to the mechanisms of these disorders.

DETAILED DESCRIPTION:
Chronic fatigue (ME/CFS) and fibromyalgia syndrome (FM) are a chronic musculoskeletal pain disorder that predominantly afflicts women. Frequently associated insomnia, cognitive abnormalities, and fatigue may lead to early disability. No consistent soft tissue abnormalities have been identified so far in these patients. The cause of these disorders is unknown, no highly effective treatment is available and the current methods of diagnosis are imprecise and unreliable. The Investigators previously used quantitative sensory testing to improve upon diagnoses of these disorders by supplementing the current procedure of manipulating defined pressure points by hand and noting the presence or absence of pain. The quantitative methods of evaluation involve repetitive application of brief, non-injurious thermal/mechanical stimulation that normally produces a moderate degree of temporal summation of sensation intensity. The patients and normal control subjects will verbally rate the magnitude of late sensations elicited by each stimulus, using a numerical scale. Chronic pain in these patients results, at least partially, from exaggerated activation of central N-methyl-D-aspartate (NMDA) receptors as a result of enhanced input from unmyelinated peripheral afferent nerve fibers supplying deep tissues. Temporal summation of second pain can lead to central sensitization with subsequent signs of hyperalgesia and allodynia. Functional brain imaging of ME/CFS and FM patients, as proposed in this study, will be used to document their ratings of repetitive experimental stimuli and the resulting pain augmentation. Successful completion of this study will provide a new method for the evaluation of chronic pain/fatigue mechanism and their response to therapy.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of FM will require a history of chronic widespread pain as well as the presence of at least eleven out of eighteen paired tender points.
* diagnosis of ME/CFS will require a history of chronic fatigue persisting or relapsing for more than 6 months as well as the presence of at least four out of eight designated symptoms.
* willing to reduce anti-depressants to low levels like amitriptyline 10 mg/day, trazodone 50 mg/day, citalopram 20 mg/day, for at least five half-lives of the medication.

Exclusion Criteria:

* Patients unwilling or unable to discontinue or modify analgesics, hypnotics, anxiolytics, or anti-depressants during the study period will be excluded from this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents living within driving distance of Gainesville, FL.
Sampling Method: Non-Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2024-10-29 (Actual)

PRIMARY OUTCOMES:
Change in experimental pain from heat pulses to the upper extremities | 3 intervals of 30 seconds each
  Numerical ratings from 0 to 100 are tied to verbal descriptors in increments of 5, to standardize the scale, and ratings in increments of 5 are permitted. Ratings of 0 and 15 designate non-painful sensations of warmth (5 = threshold for warmth, 15 = suprathreshold warmth). A rating of 20 = threshold for heat pain, 30 = very weak pain, 40 = weak pain, 50 = moderate pain, 60 = slightly strong pain, 70 = strong pain, 80 = very strong pain, 90 = extreme strong pain, and 100 = the most intense pain imaginable
Change in experimental Pain from mechanical stimulation to the upper extremities and the shoulder | 3 intervals of 30 seconds each
  Numerical ratings from 0 to 100 are tied to verbal descriptors in increments of 5, to standardize the scale, and ratings in increments of 5 are permitted. Ratings of 0 and 15 designate non-painful sensations of warmth (5 = threshold for warmth, 15 = suprathreshold warmth). A rating of 20 = threshold for heat pain, 30 = very weak pain, 40 = weak pain, 50 = moderate pain, 60 = slightly strong pain, 70 = strong pain, 80 = very strong pain, 90 = extreme strong pain, and 100 = the most intense pain imaginable

SECONDARY OUTCOMES:
Change in Fatigue Ratings | baseline and up to 3 hours.
  Visual analogue scale ratings (0-10) on a 15 cm mechanical scale. The scale is limited on the left by "no fatigue at all" and on the right by "most intense fatigue imaginable"

CONTACTS AND LOCATIONS:
Overall Officials: Roland Staud, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No